CLINICAL TRIAL: NCT04404478
Title: Stress-reduction Wellness Program for Midlife Black Women (B-SWELL)
Acronym: B-SWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Holly Jones, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-SWELL2019; K01HL141676 (NIH)
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Cardiovascular Risk Factor; Stress; Self Efficacy; Depressive Symptoms; Health Behavior
Keywords: Black women; Stress; Heart disease; Health behaviors; Midlife; Community-based research
MeSH Terms: conditions — Depression; Health Behavior; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Randomized control trial comparing intervention group (B-SWELL) with an attention control group (WE) to assess the following outcomes: healthy lifestyle scores, perceived stress scores, self efficacy, unhealthy days, and depressive symptoms.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be randomized into groups. Group sessions held online on different dates and times. Participants are asked not to share details about the study. Data collectors are blinded to participant grouping. Facilitators are blinded to the groups they are not facilitating.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-SWELL (Experimental): Participants in the B-SWELL intervention will receive information about stress and goal setting in addition to healthy lifestyle behaviors. The intervention will take place weekly for eight weeks in groups of 11 to 13 midlife Black women for peer support. Outcome measures will include perceived general health, depressive symptoms, life's simple 7 (LS7) score, and number of unhealthy days. Data collections will occur at baseline, 8 weeks, and 12 weeks.
  Interventions: Behavioral: B-SWELL: Midlife Black Women's Stress Reduction Wellness Program
- WE (Active Comparator): The attention control group (WE), will include education about healthy lifestyle behaviors and peer support. The attention control groups will also have weekly sessions for eight weeks in groups of 11 to 13 midlife Black women. Outcome measures will include perceived general health, depressive symptoms, life's simple 7 (LS7) score, and number of unhealthy days. Data collections will occur at baseline, 8 weeks, and 12 weeks.
  Interventions: Behavioral: WE: Wellness program for Midlife Black Women

INTERVENTIONS:
Behavioral: B-SWELL: Midlife Black Women's Stress Reduction Wellness Program — Stress reduction and culturally tailored information on healthy lifestyle behaviors will be used to increase healthy lifestyle behaviors according to the AHA's Life's Simple 7. Focus of intervention on per support, goal setting, stress reduction, and culturally relevant information.
  Arms: B-SWELL
Behavioral: WE: Wellness program for Midlife Black Women — Culturally tailored information will be provided about healthy lifestyle behaviors will be used to increase healthy lifestyle behaviors according to the AHA's Life's Simple 7. Focus of intervention on peer support and culturally relevant content.
  Arms: WE

SUMMARY:
This research study examines the unique cultural and gender-based factors that influence how midlife Black women experience stress and incorporate healthy lifestyle behaviors into daily life. The B-SWELL intervention uses stress reduction and goal setting to increase self efficacy in adopting healthy lifestyle behaviors. The B-SWELL intervention will be compared to an inattention control wellness group in a randomized control trial. The long-term outcome is to decrease cardiovascular disease risk in this high-risk population, midlife Black women.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the primary cause of death in all women, and as women transition through midlife, the prevalence of CVD exceeds that of men.1 Midlife Black women, defined as ages 40-64,unduly shoulder the burden of CVD (49%), hypertension (40%), and heart failure (50% greater risk). Midlife Black women also report higher levels of chronic stress and greater numbers of stressful life events in comparison to midlife White women, putting them at greater risk for CVD. In addition to the physical impact, coping with chronic stress takes time and energy away from self-care, functioning as a barrier to the adoption of healthy lifestyle behaviors. Existent interventions do not fully address the unique factors contributing to the experience of stress, lifestyle behaviors, and CVD risk in midlife Black women.

The purpose of this research proposal is to develop a midlife Black women's Stress-reduction WELLness intervention, B-SWELL, to promote healthy lifestyle behaviors based on the stressors and themes identified in preliminary research. Community-based participatory research (CBPR) methods will be used to engage the community and include midlife Black women in the development of the B-SWELL. We propose that the skills and knowledge gained through participation in the B-SWELL program will increase receptivity to the healthy lifestyle behaviors outlined in the American Heart Association's Life Simple 7 Success Plan (LS7). The LS7 targets seven risk factors known to increase cardiovascular related health risk: cholesterol, fasting glucose, blood pressure, body mass index, physical activity, diet, and smoking.

Our hypothesis proposes that low stress scores and greater self efficacy will be associated with the adoption of AHA's healthy lifestyle behaviors. Low stress and self efficacy will be facilitated through peer support and culturally relevant content, materials, and themes. B-SWELL participants will show improved self-efficacy in managing life stress and adopting the LS7 behaviors, compared to a control group receiving traditional wellness education (WE group).

Aim 1: Develop the B-SWELL intervention for midlife Black women through the innovative leveraging of CBPR methodology and LS7 modifiable healthy lifestyle behaviors.

1. To develop components of the B-SWELL intervention prototype for midlife Black women.
2. Obtain ratings of the new components of the B-SWELL from our community advisory board for degree of accuracy, relevance, and feasibility to inform further refinements.

Aim 2: Determine the feasibility of the B-SWELL intervention with a trial of 50 midlife Black women randomized to the B-SWELL intervention (25) or to a wellness education (WE) control group (25):

1. Obtain recruitment, retention, treatment fidelity ratings, and satisfaction ratings for the intervention procedures for both groups;
2. Compare mediator measures (stress, self-efficacy) for participants in the B-SWELL intervention group with those in the WE group at 8 and 12 weeks.
3. Compare outcome measures (LS7 summary scores, unhealthy days, general health, depressive symptoms) for participants in the B-SWELL intervention group with those in the WE attention control group at 8 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* fluent in the English language,
* ability to hear and talk well enough to engage in everyday conversation,
* access to a telephone with messaging,
* access to WIFI,
* willingness to participate for duration of the study.

Exclusion Criteria:

* recent immigration to the U.S.,
* prisoner or on house arrest,
* pregnant,
* terminal illness (i.e., late stage cancer, end-of-life condition, renal failure requiring dialysis),
* history of Alzheimer's, dementia, or severe mental illness (i.e., suicidal tendencies, schizophrenia, or severe untreated depression),
* any other major health conditions or disabilities prohibiting safe participation in the program.

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Midlife Black/African-American women between the ages of 40 and 64,
Enrollment: 52 (Actual)
Dates: Start 2021-02-13 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly J Jones, PhD,RN,NP, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, College of Nursing, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We anticipate that there will be manuscripts, not only from the findings addressing Specific Aims 1 and 2, but also from secondary analyses from data generated from this study. We will disseminate results from Specific Aims 1 and 2, as well as results from secondary analyses, in peer-reviewed journals. We will also make the data available to others. Data will be shared with undergraduate honors students, MSN students, DNP students, PhD students, post-doctoral students, and interested faculty members at the University of Cincinnati, College of Nursing, and other institutions.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available upon completion of the study and remain available for 1 year.
Access Criteria: To be determined.

REFERENCES:
- [Background] Jones HJ, Norwood CR, Bankston K. Leveraging Community Engagement to Develop Culturally Tailored Stress Management Interventions in Midlife Black Women. J Psychosoc Nurs Ment Health Serv. 2019 Mar 1;57(3):32-38. doi: 10.3928/02793695-20180925-01. Epub 2018 Oct 1. PMID 30272812
- [Background] Jones HJ, Norwood CR, Bankston K, Bakas T. Stress Reduction Strategies Used by Midlife Black Women to Target Cardiovascular Risk. J Cardiovasc Nurs. 2019 Nov/Dec;34(6):483-490. doi: 10.1097/JCN.0000000000000615. PMID 31609281
- [Background] Jones HJ, Sternberg RM, Janson SL, Lee KA. A Qualitative Understanding of Midlife Sources of Stress and Support in African-American Women. J Natl Black Nurses Assoc. 2016 Jul;27(1):24-30. PMID 29932540
- [Background] Jones HJ, Bakas T, Nared S, Humphries J, Wijesooriya J, Butsch Kovacic M. Co-Designing a Program to Lower Cardiovascular Disease Risk in Midlife Black Women. Int J Environ Res Public Health. 2022 Jan 26;19(3):1356. doi: 10.3390/ijerph19031356. PMID 35162379
- [Background] Jones HJ, Kovacic MB, Bakas T. Establishing Validity of the Midlife Black Women's Stress-Reduction Wellness Program Materials Using a Mixed Methods Approach. J Cardiovasc Nurs. 2022 Sep-Oct 01;37(5):446-455. doi: 10.1097/JCN.0000000000000876. Epub 2021 Dec 22. PMID 34935740
- [Derived] Jones HJ, Kovacic MB, Bacchus P, Almallah W, Bakas T. Participant Satisfaction in a Cardiovascular Disease Prevention Intervention for Midlife Black Women. West J Nurs Res. 2024 Jan;46(1):3-9. doi: 10.1177/01939459231208420. Epub 2023 Oct 31. PMID 37905540
- [Derived] Jones HJ, Butsch Kovacic M, Lambert J, Almallah WR, Becker R, de las Fuentes L, Bakas T. A randomized feasibility trial of the Midlife Black Women's Stress and Wellness intervention (B-SWELL); a community participatory intervention to increase adoption of Life's Simple 7 healthy lifestyle behaviors. Transl Behav Med. 2022 Nov 21;12(11):1084-1095. doi: 10.1093/tbm/ibac075. PMID 36208220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from the community using fliers, social media, email list serves, and word of mouth. The recruitment efforts were led by community partners. Recruitment was completed within 7 weeks.
Pre-assignment Details: Of the 52 persons randomized and enrolled in the study, 3 persons withdrew prior to the start of the study (week 1) and 1 person was withdrawn prior to week 2 for lack of participation.
Groups:
- B-SWELL Intervention Group (B-SWELL): Black women's stress and wellness intervention
- Wellness (WE): Comparison group
Period: Overall Study
Arm/Group | B-SWELL Intervention Group (B-SWELL) | Wellness (WE)
Started | 26 | 26
Completed | 25 | 23
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- B-SWELL Group: The Midlife Black women's Stress and Wellness group (B-SWELL) is the intervention group.
- WE Group: The Wellness (WE) group is the comparison group.
- Total: Total of all reporting groups
Arm/Group | B-SWELL Group | WE Group | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Customized [Number; unit: participants] — midlife Black women were recruited between the ages of 40 and 64. Age was self reported using month and birth year.
  participants
    Age between 40 and 64 | 25 | 23 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 23 | 48
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: American Heart Association's Life's Simple Seven (LS7) Score
Description: Life's Simple 7 score measures cardiovascular health. Minimum score is 0. Maximum score is 14. Each of the 7 metrics (weight loss, diet, exercise, cholesterol management, glucose management, smoking, and blood pressure management) is rated 0 (poor), 1 (average), or 2 (best). Higher scores indicate greater cardiovascular health. Lower scores indicate greater risk for heart disease.
Time Frame: Baseline to 12 weeks
Population: These measures were used to calculate the differences between timepoints for the two groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- WE (Wellness Comparison Group): The attention control group (WE), will include education about healthy lifestyle behaviors and peer support. The attention control groups will also have weekly sessions for eight weeks in groups of 11 to 13 midlife Black women. Outcome measures will include perceived general health, depressive symptoms, life's simple 7 (LS7) score, and number of unhealthy days. Data collections will occur at baseline, 8 weeks, and 12 weeks.
  WE: Wellness program for Midlife Black Women: Culturally tailored information will be provided about healthy lifestyle behaviors will be used to increase healthy lifestyle behaviors according to the AHA's Life's Simple 7. Focus of intervention on peer support and culturally relevant content.
Arm/Group | B-SWELL | WE (Wellness Comparison Group)
Number analyzed (Participants) | 25 | 23
units on a scale | 8.76 (2.11) | 8.21 (2.50)

2. Secondary Outcome: Unhealthy Days
Description: 'Unhealthy Days' is measures by the number of unhealthy days reported by the participant. This question asks the participant how many days in past month that their physical/mental health was not good. This is a continuous numeric response. Higher numbers indicate poorer health during the reported timeframe.
Time Frame: baseline to 12 weeks
Population: The number of unhealthy days measured within 2 weeks.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | B-SWELL | WE (Wellness Comparison Group)
Number analyzed (Participants) | 25 | 23
days | 2.52 (6.26) | 3.09 (4.86)

3. Secondary Outcome: Perceived General Health
Description: The Perceived General Health question is one item from the Short Form Health Survey. The participants will rate their health as 'excellent', 'very good', 'good', 'fair' and 'poor'. Responses are categorical. The reported outcome reflects the number of participants who rate their health as 'good'.
Time Frame: Baseline to 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- B-SWELL: Intervention group
- WE - Wellness Group: comparison group
Arm/Group | B-SWELL | WE - Wellness Group
Number analyzed (Participants) | 25 | 23
Participants | 17 | 13

4. Secondary Outcome: Patient Health Questionnaire (PHQ9)
Description: The PHQ9 measures depressive symptoms. Participants rate their depressive symptoms from '0' (not at all) to '3' (every day). Scores range from 0 to 27. Higher scores indicate greater risk of clinical depression. Lower scores indicate less risk for depression.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B-SWELL | WE - Wellness Group
Number analyzed (Participants) | 25 | 23
units on a scale | 4.80 (5.17) | 5.39 (3.20)

5. Other Pre Specified Outcome: Cohen's Perceived Stress Scale (PSS-10)
Description: The Perceived stress scale (PSS-10) measures a person's perception of general stress. Items are rated on a scale of 0 to 4 with a maximum score of 40. Higher levels of stress correspond with higher scores. Low scores indicate less stress.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B-SWELL | WE - Wellness Group
Number analyzed (Participants) | 25 | 23
units on a scale | 16.68 (6.32) | 15.39 (5.48)

6. Other Pre Specified Outcome: General Self-Efficacy Scale (GSE)
Description: The GSE is a 10-item psychometric scale that assesses optimistic self-beliefs to cope with life demands. The total score is calculated by finding the sum of the all items. Scores range from 1 (not at all true) to 4 (exactly true). Total scores range between 10 and 40. A higher score indicates greater self-efficacy in achieving a particular outcome. Lower scores indicate the participant has less self-efficacy in achieving the outcome.
Time Frame: baseline to 12 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B-SWELL | WE - Wellness Group
Number analyzed (Participants) | 25 | 23
units on a scale | 33.44 (3.36) | 32.91 (2.70)

7. Other Pre Specified Outcome: Satisfaction (Adapted From Satisfaction Questionnaire).
Description: Satisfaction. Participants rate their satisfaction of the overall B-SWELL program using a Likert type scale ranging from 1=strongly disagree to 5=strongly agree. The questionnaire includes items for usefulness, ease of use, and acceptability of the intervention. Ratings are averaged across participants.
  The results reported here refer to the question: 'The weekly program materials addressed the problems I was having as a midlife Black woman.'
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B-SWELL | WE - Wellness Group
Number analyzed (Participants) | 25 | 23
units on a scale | 4.52 (0.92) | 4.30 (0.70)

ADVERSE EVENTS:
Time Frame: 12 weeks: Time point 1 (0 weeks), Time point 2 ( 8 weeks), and Timepoint 3 (12 weeks)
Arm/Group | B-SWELL | WE - Wellness Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

LIMITATIONS AND CAVEATS:
Limitations include:

* The comparison group included culturally tailored materials and was not a true control.
* The effects of peer support and group interactions may have been underestimated in the WE group.
* The threat of group contamination could not be eliminated.
* The small sample in this feasibility study prohibits our ability to make inferences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT04404478/Prot_SAP_000.pdf